CLINICAL TRIAL: NCT02380898
Title: Preemptive Ketorolac for Intraoperative Shoulder Tip Pain During Cesarean Section: A Double-Blind Randomized Clinical Trial.
Brief Title: Preemptive Ketorolac for Shoulder Tip Pain During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, lecturer of anesthesia and ICU, Assiut University,Assiut, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ketorolac
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2015-12

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Ketorolac; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ketorolac (Experimental)
  Interventions: Drug: Ketorolac
- Normal saline 0.9% (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketorolac — 30 mg ketorolac immediately before induction of anesthesia
  Arms: Ketorolac
Drug: Normal saline — 4 mL normal saline 0.9% immediately before induction of anesthesia
  Arms: Normal saline 0.9%

SUMMARY:
Our study is planned to investigate if pre-emptive Ketorolac would decrease the incidence of intraoperative shoulder tip pain and improve discomfort during Caesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is the most frequent major abdominal surgery among women worldwide . Shoulder pain, is a common but mostly neglected consequence of caesarean section and little is known about this entity. The pain is described as sharp, deep and referred, usually begins intraoperatively and continue for 2-3 days after surgery.

Although infant and maternal death rates have been decreased after CS, this procedure is not free of risks for mother and child. Compared with normal vaginal delivery (NVD), some CS complications include: more haemorrhage; increased postoperative pain; atelectasia; nausea; vomiting; risks for wound infection or wound opening and shoulder pain.

Although spinal anaesthesia (SA) is a common technique for CS in the past decade, and there are many studies about CS complications, there are few studies about shoulder pain as one of CS complications. Kikuchi et al. reported that women undergoing cesarean section under compined spinal epidural anaethesia experience shoulder-tip pain with great frequency. Our study was planned and performed to investigate if pre-emptive Ketorolac would decrease the incidence of intraoperative shoulder pain and improve discomfort during CS.

Sharp pain observed in these patients was experienced in the shoulder area or under the diaphragm. The pain was described as coming from deep within the shoulder, and in some, would seem to radiate from the right chest. The pain spread down the upper right arm and up the right neck in some, resulting in muscular tension and pain. The cause of this pain is postulated to sub-diaphragmatic air trapping, subdiaphragmatic clot or peritoneal irritation. This type of shoulder pain is reported commonly after laparoscopic surgery and it is reported that heat, massage and drinking hot water or hot tea with fresh lemon relieves this pain.

ELIGIBILITY:
Inclusion Criteria:

* nulligravida healthy women who delivered single term baby, with American Society of Anesthesiologists physical status 1 or 2

Exclusion Criteria:

previous caesarean section; pre-eclampsia; gestational diabetes; trauma; fractures or chronic pain in shoulder joints, forearms, upper limbs; cardiovascular or biliary system disorders; women undergoing emergency caesarean; previous history of abdominal surgery; conditions preventing spinal block, including local infection; coagulopathies; haemodynamic instability

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Intraoperative shoulder tip pain | intraoperative

SECONDARY OUTCOMES:
pain score VAS | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt

REFERENCES:
- [Derived] Abbas MS, Askar OA, Abdel Aleem AA. Pre-emptive ketorolac for prevention of intraoperative shoulder pain in patients undergoing cesarean section: A double blind randomized clinical trial. Asian J Anesthesiol. 2017 Sep;55(3):68-72. doi: 10.1016/j.aja.2017.07.002. Epub 2017 Sep 20. PMID 28993164